CLINICAL TRIAL: NCT02316704
Title: Fixation of OsseoTi™ Porous Structure Versus PPS (Porous Plasma Spray) Coating on the G7™ Acetabular Component for Primary Total Hip Arthroplasty: A Single-Blinded Randomized Controlled Trial Evaluating Implant Migration, Acetabular Liner Wear, and Patient Reported Outcome
Brief Title: Fixation of OsseoTi™ Porous Structure Versus PPS (Porous Plasma Spray) Coating on the G7™ Acetabular Component for Primary Total Hip Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirill Gromov, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G7_RSA_v1.02
Record Dates: First submitted 2014-12-06; First posted 2014-12-15 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- OsseoTi™ G7 large (Active Comparator): OsseoTi™ G7 acetabular cup and an E1™ liner holding largest possible femoral head (36mm-44mm)
  Interventions: Device: THA with G7 PPS coted acetabular component; Device: THA with G7 OsseoTi coted acetabular component
- OsseoTi™ G7 32 (Active Comparator): OsseoTi™ G7 acetabular cup and an E1™ insert holding a 32mm femoral head
  Interventions: Device: THA with G7 PPS coted acetabular component; Device: THA with G7 OsseoTi coted acetabular component
- conventional PPS coated G7 large (Active Comparator): conventional PPS coated G7 acetabular cup and an E1™ insert holding largest possible femoral head (36mm-44mm)
  Interventions: Device: THA with G7 PPS coted acetabular component; Device: THA with G7 OsseoTi coted acetabular component
- conventional PPS coated G7 32 (Active Comparator): conventional PPS coated G7 acetabular cup and an E1™ insert holding a 32mm femoral head
  Interventions: Device: THA with G7 PPS coted acetabular component; Device: THA with G7 OsseoTi coted acetabular component

INTERVENTIONS:
Device: THA with G7 PPS coted acetabular component
Device: THA with G7 OsseoTi coted acetabular component

SUMMARY:
The primary objective of this project is to investigate, using RSA, acetabular implant migration of the OsseoTi™ G7 acetabular cup in comparison to conventional PPS coated G7 acetabular cup, and compare liner wear of thinnest available E1™ liner, allowing for the largest possible femoral head (36mm-44mm) to E1™ liner holding a 32mm femoral head in the G7 acetabular system with endpoint assessment being performed at the 2 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* • Participants with primary hip osteoarthritis set to receive a primary unilateral uncemented total hip arthroplasty.

  * Participants must be 18-75 years of age.
  * Participants must be able to speak and understand Danish (or depending on country where patient is enrolled).
  * Participants must be able to give informed consent and be cognitively intact.
  * Participants must be expected to be able to complete all postoperative controls.
  * Participants must not have severe comorbidities, ASA-score ≤ 3.

Exclusion Criteria:

* Terminal illness.
* Rheumatoid arthritis.
* Previous fracture of the hip.
* Osteonecrosis of the hip.
* Previous infection of the hip.
* Severe bony deformity warranting the use of non-standard implants.
* Metastasis in the periarticular bone or proximal femur.
* Female patients that are pregnant or planning pregnancy during follow-up period
* If bone stock or femoral canal type, assessed on preoperative x-ray, warrants the use of cemented fixation.
* Documented osteoporosis with patient in active medical treatment.
* Comorbidity with altered pain perception (e.g. DM with neuropathy).
* Participants that develop deep infection in the follow-up period are excluded from the project.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
RSA migration in 3 dimentions of the acetabular components as measured by Radiostereometric analysis, RSA. | 2 year
  Radiostereometric analysis, RSA, is an accurate technique for measuring small relative motions from sequential sets of radiographs over time and has been used to measure polyethylene wear and implant migration. Measurements are performed in microns.

CONTACTS AND LOCATIONS:
Locations (2):
- Dept. of Orthopaedic Surgery, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark
- Sahlgrenska University Hospital, Department of Orthopedics,, Gothenburg, Sweden